CLINICAL TRIAL: NCT03987490
Title: A Feasibility Trial of Parent-targeted Strategies to Increase HPV Vaccination
Brief Title: Usability of HPV Vaccine Reminders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: IRB201500997
Record Dates: First submitted 2019-06-11; First posted 2019-06-17 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Human Papilloma Virus (HPV)
Keywords: vaccine
MeSH Terms: interventions — Standard of Care; Motivational Interviewing

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parents of Girls (Experimental): Parents of 11-to-12-year-old girls who did not have records of the HPV vaccine in the EHR or Medicaid claims.
  Interventions: Behavioral: Text Message; Behavioral: Standard of Care; Behavioral: Motivational Interview
- Parents of Boys (Experimental): Parents of 11-to-12-year-old girls who did not have records of the HPV vaccine in the EHR or Medicaid claims.
  Interventions: Behavioral: Text Message; Behavioral: PostCard; Behavioral: Standard of Care; Behavioral: Motivational Interview

INTERVENTIONS:
Behavioral: Text Message — Vaccine reminder notification sent via text
Behavioral: PostCard — Vaccine reminder notification sent via standard mail
  Arms: Parents of Boys
Behavioral: Standard of Care — No additional information given to parents
Behavioral: Motivational Interview — Phone-based semi-guided discussion with parents who had not yet agreed to vaccination after reminders sent

SUMMARY:
This study will assess the usefulness of parent-targeted strategies in improving care seeking among parents of 11-12 year old adolescents. Specifically, the study team will focus on reminders (postcard or text message) and motivational interviewing to improve adolescent vaccination.

DETAILED DESCRIPTION:
Despite the impressive cancer preventing potential of human papillomavirus (HPV) vaccines, HPV vaccine coverage rates in the United States remain substantially lower than other vaccines and Healthy People 2020 targets. HPV vaccine initiation can be improved through targeted reminders that motivate parents. Our long-term goal is to maximize HPV vaccination rates among girls and boys within the United States using efficient and sustainable strategies. The objective of this protocol is to evaluate the usefulness of a tiered strategy of a parent-targeted strategies in improving care seeking and receptiveness to vaccine recommendations. Strategies include HPV vaccine reminders via postcard or text message and phone-based Motivational Interview sessions. The central hypothesis is addressing key health beliefs (e.g., perceived benefits and barriers) will increase parental acceptance and, thus, HPV vaccine initiation.

ELIGIBILITY:
Inclusion Criteria:

* Parents of 11-12 year olds who attend the Schiebler CMS clinic at University of Florida in the previous year

Exclusion Criteria:

* Unable to meet inclusion criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2016-12-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients with deliverable text messages | up to 2 weeks
  Percentage of Patients with deliverable text messages
Percentage of phone calls where interviewer is adherent to MI | During phone interview
  Adherence to MI

SECONDARY OUTCOMES:
Percentage of adolescent who get one dose of the HPV vaccine | Six months
  HPV vaccine initiation (1 dose)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Staras, Principal Investigator — University of Florida
Locations (1):
- UF Health Pediatrics - Gerold L. Schiebler CMS Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No